CLINICAL TRIAL: NCT06901557
Title: Benefits of Jing-Si-Herbal-Tea in Bronchiectasis
Acronym: JSHT-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Chou-Chin Lan, Head of Division of Pulmonary Medicine, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-XD-053
Record Dates: First submitted 2024-09-09; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: Patients are divided into two groups: the usual care group (UC group) and the Jing-Si Herbal Tea group (JSHT group).
  The UC group will receive standard medical treatment, with one placebo packet daily for three months.
  The JSHT group will receive the standard medical treatment along with Jing-Si Herbal Tea, one packet daily for three months.
  There were 12 participants in JSHT group and thirteen in UC group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- usual care group (UC group) (Placebo Comparator): The UC group will receive standard medical treatment, with one placebo packet daily for three months.
  Interventions: Combination Product: Placebo
- Jing-Si Herbal Tea group (JSHT group) (Experimental): The JSHT group will receive the standard medical treatment along with Jing-Si Herbal Tea, one packet daily for three months.
  Interventions: Combination Product: Jing-Si Herbal Tea

INTERVENTIONS:
Combination Product: Jing-Si Herbal Tea — The JSHT group will receive the standard medical treatment along with Jing-Si Herbal Tea, one packet daily for three months.
  Arms: Jing-Si Herbal Tea group (JSHT group)
Combination Product: Placebo — The UC group will receive standard medical treatment, with one placebo packet daily for three months.
  Arms: usual care group (UC group)

SUMMARY:
Patients are divided into two groups: the usual care group (UC group) and the Jing-Si Herbal Tea group (JSHT group).

* **UC Group**: Receives standard treatment and one placebo packet daily for three months.
* **JSHT Group**: Receives standard treatment plus one packet of Jing-Si Herbal Tea daily for three months.

Each group includes 30 participants. The study runs from January 1, 2014, to December 31, 2014. Exclusions include severe liver or renal dysfunction and allergy to Jing-Si Herbal Tea. Participants must follow the study protocol.

**Assessments**:

* **HRQL**: Measured using the COPD Assessment Test (CAT) and the Modified Medical Research Council (mMRC) scale.
* **Blood Tests**: Include WBCs, hemoglobin, hematocrit, platelets, BUN, creatinine, uric acid, liver enzymes, electrolytes, CRP, and pPro-BNP. Blood samples will also be analyzed for DAMPs and inflammatory cytokines.
* **Pulmonary Function Tests (PFT)**: Conducted with a spirometer per American Thoracic Society guidelines.

DETAILED DESCRIPTION:
Patients are divided into two groups: the usual care group (UC group) and the Jing-Si Herbal Tea group (JSHT group).

The UC group will receive standard medical treatment, with one placebo packet daily for three months.

The JSHT group will receive the standard medical treatment along with Jing-Si Herbal Tea, one packet daily for three months.

Each group will enroll 30 participants. Study period: From January 1, 2014, to December 31, 2014. During the study, participants with contraindications such as severe liver dysfunction, severe renal dysfunction, or a history of allergy to JSHT are excluded from enrollment based on the exclusion criteria at the time of enrollment. The only requirement for participants is to adhere to the study protocol regarding the consumption of JSHT and undergoing tests.

Baseline and post-treatment HRQL were assessed using the COPD assessment test (CAT), along with blood tests including white blood cells (WBCs), percentages of different types of WBCs (neutrophils, lymphocytes, monocytes, eosinophils, basophils), hemoglobin (Hb), hematocrit (Hct), platelets (PLT), blood urea nitrogen (BUN), creatinine (Cr), uric acid (UA), liver enzymes (aspartate aminotransferase, alanine aminotransferase), electrolytes (sodium, potassium), C-reactive protein (CRP), and pro-brain natriuretic peptide (pPro-BNP). Blood samples from patients will be analyzed for DAMPs and inflammatory cytokines.

Health-related quality of life (HRQL) The Taiwan Society of Pulmonary and Critical Care Medicine offers the Chinese version of the COPD Assessment Test (CAT) on the website. This test consists of eight items designed to evaluate COPD symptoms. These symptoms include cough, phlegm production, chest tightness, breathlessness, limitations in daily activities, confidence in leaving the house, sleep disturbances, and energy levels. Each symptom is rated on a scale from 0 to 5, culminating in a total CAT score ranging from 0 to 40. A higher score reflects more severe COPD symptoms. A score of 10 or higher is indicative of a significant symptom burden. The Modified Medical Research Council (mMRC) scale was used to evaluate dyspnea. This scale, comprising a 5-point grading system ranging from 0 to 4, measures dyspnea severity. A score of 0 indicates dyspnea only during intense exercise, while a sore of 4 represents breathlessness at rest.

Pulmonary function tests (PFT) PFT were conducted using a spirometer following the guidelines set by the American Thoracic Society.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Clinically diagnosed with bronchiectasis
3. Willing to participate in the study
4. Signed an informed consent form

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Individuals with severe liver
3. Individuals with severe kidney diseases
4. Individuals who refuse to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQL) | The HRQL will be assessed at baseline and after three months of intervention.
  The Taiwan Society of Pulmonary and Critical Care Medicine offers the Chinese version of the COPD Assessment Test (CAT) on the website. This test consists of eight items designed to evaluate COPD symptoms. These symptoms include cough, phlegm production, chest tightness, breathlessness, limitations in daily activities, confidence in leaving the house, sleep disturbances, and energy levels. Each symptom is rated on a scale from 0 to 5, culminating in a total CAT score ranging from 0 to 40. A higher score reflects more severe COPD symptoms. A score of 10 or higher is indicative of a significant symptom burden. The Modified Medical Research Council (mMRC) scale was used to evaluate dyspnea. This scale, comprising a 5-point grading system ranging from 0 to 4, measures dyspnea severity. A score of 0 indicates dyspnea only during intense exercise, while a sore of 4 represents breathlessness at rest.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Xindan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The investigators have decided not to share individual participant data (IPD) due to several important considerations. Protecting participant privacy is our top priority, as sharing IPD could expose sensitive personal information and pose risks of re-identification, even if de-identified. Additionally, participants did not consent to their data being shared with other researchers, and obtaining re-consent would be challenging. Ensuring data security also requires significant resources and technical measures that our current infrastructure may not support. Furthermore, complying with complex legal and ethical regulations surrounding data sharing adds another layer of complexity. Finally, maintaining the quality and integrity of IPD before sharing demands extra effort and resources. These factors collectively influence our decision to prioritize participant protection and data security.

REFERENCES:
- [Background] Kao SW, Chang YC, Lin FH, Huang TL, Chen TS, Lin SZ, Lin KH, Kuo WW, Ho TJ, Huang CY. Jing-Si Herbal Tea Suppresses H2O2 -Instigated Inflammation and Apoptosis by Inhibiting Bax and Mitochondrial Cytochrome C Release in HIG-82 Synoviocytes. Environ Toxicol. 2024 Dec;39(12):5347-5356. doi: 10.1002/tox.24406. Epub 2024 Sep 5. PMID 39234996
- [Background] Lin HC, Hsieh MH, Lo YL, Huang HY, Huang SW, Huang CD, Chang PJ, Lo CY, Lin TY, Fang YF, Lin SM, Lin CY, Tsai YH. IL-6 and TIMP-1 Correlated to Airway Pathogen Colonization and Predict Disease Severity in Patients with Non-Cystic Fibrosis Bronchiectasis. J Inflamm Res. 2024 Aug 28;17:5701-5709. doi: 10.2147/JIR.S465413. eCollection 2024. PMID 39219819